CLINICAL TRIAL: NCT00105547
Title: Phase 3, Multicenter, Randomized, Double Blind, Placebo Controlled Study of the Effect of Daily Treatment With MPC-7869 on Measures of Cognition, Activities of Daily Living and Global Function in Subjects With Mild Dementia of the Alzheimer's Type
Brief Title: Efficacy Study of MPC-7869 to Treat Patients With Alzheimer's
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Ed Swabb, MD, Myriad Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MPC-7869-04-005.02
Record Dates: First submitted 2005-03-15; First posted 2005-03-16 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Alzheimer's; Dementia; Dementia of Alzheimer Type
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — tarenflurbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 800 mg BID
  Interventions: Drug: MPC-7869
- 2 (Placebo Comparator): BID dosing
  Interventions: Drug: MPC-7869

INTERVENTIONS:
Drug: MPC-7869 — oral 800 mg BID
  Arms: 1
Drug: MPC-7869 — Oral BID dosing
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the change in cognitive ability and activities of daily living in patients with Alzheimer's disease (AD) as measured by specific evaluations during 18 months of dosing.

DETAILED DESCRIPTION:
This trial is a phase 3, multicenter, randomized, double-blind, placebo controlled, parallel group study comparing the safety and efficacy of daily dosing of MPC-7869 to placebo. The study subjects will have the diagnosis of mild dementia of the Alzheimer's type. Subjects may be taking approved medication for Alzheimer's disease provided the dose has been stable for at least 6 months.

The primary objective of the study is to evaluate the change in cognition and activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Have had a diagnosis of probable Alzheimer's disease.
* Men or women ages 55 years or greater and living in the community at the time of enrollment (i.e., not living in a rest home or nursing care facility).
* Signed the subject Informed Consent Form and is willing and able to participate for the duration of the study.
* Ability to read and understand English or Spanish to ensure compliance with cognitive testing and study visit procedures.
* Female subjects must be surgically sterile or postmenopausal for > 1 year.
* Subjects currently taking approved medication for Alzheimer's disease for at least six months prior to day 1 may be enrolled.
* Subjects must have a reliable caregiver who can read, understand and speak English or Spanish.

Exclusion Criteria:

* Current evidence of other causes of dementia.
* History or evidence of, active malignancy, except for basal cell carcinoma or squamous cell carcinoma of the skin, within the 24 months prior to entry. Men with prostate cancer may be enrolled at the discretion of the sponsor.
* Chronic or acute renal, hepatic or metabolic disorder.
* Use of any investigational therapy within 30 days, or 5 half-lives, whichever is longer, and/or use of AD immunotherapy prior to screening.
* Major surgery and related complications not resolved within 12 weeks prior to Day 1.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2005-02; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Cognition and activities of daily living | 18 mos

SECONDARY OUTCOMES:
Global function and behavior | 18 mos

CONTACTS AND LOCATIONS:
Overall Officials: Ed Swabb, MD, Study Director — Myrexis Inc.
Locations (114):
- United States (114):
  - Alabaster, Alabama
  - Huntsville, Alabama
  - Mesa, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Sun City, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Fresno, California
  - Irvine, California
  - La Jolla, California
  - Lafayette, California
  - Laguna Hills, California
  - Long Beach, California
  - Los Angeles, California
  - Newport Beach, California
  - Oceanside, California
  - Rancho Mirage, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Vista, California
  - Denver, Colorado
  - Danbury, Connecticut
  - Darien, Connecticut
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Bay Harbor, Florida
  - Boca Raton, Florida
  - Clearwater, Florida
  - Derrfield Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Naples, Florida
  - North Miami, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Plantation, Florida
  - Pompano Beach, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Chicago, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Glen Burnie, Maryland
  - Boston, Massachusetts
  - Brockton, Massachusetts
  - West Yarmouth, Massachusetts
  - Farmington Hills, Michigan
  - Grand Rapids, Michigan
  - Rochester, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Kenilworth, New Jersey
  - Morristown, New Jersey
  - Piscataway, New Jersey
  - Princeton, New Jersey
  - Stratford, New Jersey
  - Toms River, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - Elmsford, New York
  - New York, New York
  - Olean, New York
  - Rochester, New York
  - Syracuse, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Centerville, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Jenkintown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Scotland, Pennsylvania
  - East Providence, Rhode Island
  - Providence, Rhode Island
  - Beaufort, South Carolina
  - Greer, South Carolina
  - North Charleston, South Carolina
  - Johnson City, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Galveston, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Wichita Falls, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Bennington, Vermont
  - Alexandria, Virginia
  - Charlottesville, Virginia
  - Virginia Beach, Virginia
  - Middleton, Wisconsin
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Green RC, Schneider LS, Amato DA, Beelen AP, Wilcock G, Swabb EA, Zavitz KH; Tarenflurbil Phase 3 Study Group. Effect of tarenflurbil on cognitive decline and activities of daily living in patients with mild Alzheimer disease: a randomized controlled trial. JAMA. 2009 Dec 16;302(23):2557-64. doi: 10.1001/jama.2009.1866. PMID 20009055